CLINICAL TRIAL: NCT04541225
Title: Phase 1/2 Dose Escalation, Safety, Pharmacokinetics, and Efficacy Study of NUV-422 in Adults With Recurrent or Refractory High-grade Gliomas and Solid Tumors
Brief Title: Study of NUV-422 in Adults With Recurrent or Refractory High-grade Gliomas and Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Nuvation Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NUV-422-02
Record Dates: First submitted 2020-08-21; First posted 2020-09-09 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Glioma; Glioma, Malignant; Glioma, Mixed; Glial Cell Tumors; Breast Cancer; Breast Carcinoma; Cancer of Breast; Cancer of the Breast; Breast Tumor; Malignant Tumor of Breast; Advanced Breast Cancer; Advanced Breast Carcinoma; Metastatic Breast Cancer; Metastatic Breast Carcinoma; Prostate Cancer; Prostatic Cancer; Cancer of Prostate; Cancer of the Prostate; Prostate Neoplasm; Castrate Resistant Prostate Cancer; Castration-resistant Prostate Cancer; Castration Resistant Prostatic Neoplasms; Glioblastoma; Recurrent Glioblastoma
Keywords: Phase 1; malignant glioma; metastatic breast cancer; metastatic castration-resistant prostate cancer
MeSH Terms: conditions — Glioma; Breast Neoplasms; Prostatic Neoplasms; Prostatic Neoplasms, Castration-Resistant; Glioblastoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Phase 1 Dose Escalation (Experimental): NUV-422 will be administered at escalating dose levels until the maximum tolerated dose (MTD) is reached.
  Interventions: Drug: NUV-422

INTERVENTIONS:
Drug: NUV-422 — NUV-422 is an investigational drug for oral dosing.

SUMMARY:
At the time of study termination, NUV-422-02 was a first-in-human, open-label, Phase 1 dose escalation study designed to evaluate the safety and efficacy of NUV-422. The study population comprised adults with recurrent or refractory high-grade gliomas (HGGs), metastatic breast cancer (mBC), with and without brain metastases, and recurrent or refractory metastatic castration-resistant prostate cancer (mCRPC). All patients self-administered NUV-422 orally in 28-day cycles until disease progression, toxicity, withdrawal of consent, or termination of the study.

ELIGIBILITY:
Key Inclusion Criteria

For All Cohorts:

1. Recovered from toxicity to prior anti-cancer therapy
2. Adequate bone marrow and organ function
3. Appropriate candidate for NUV-422 monotherapy
4. Life expectancy of > 3 months

Cohort-Specific Inclusion Criteria: In addition to the inclusion criteria listed above, the following criteria apply based on enrollment into specific cohorts.

High-Grade Glioma:

1. Histologically confirmed diagnosis of high-grade glioma
2. Evidence of recurrence after treatment (ie, surgery, radiation, or temozolomide) or refractory (or intolerant) to treatment
3. Measurable or non-measurable disease
4. Karnofsky Performance Status (KPS) score ≥ 60

HR+HER2- Metastatic Breast Cancer:

1. Men and women who are not suitable for surgical resection or radiotherapy for the purpose of cure
2. Diagnosis of locally advanced or HR+HER2- metastatic breast cancer
3. Evidence of progression as determined by the Investigator per standard criteria
4. Patients must have endocrine-resistant disease
5. Prior therapy: At least 1 but not more than 4 prior lines of systemic therapies for locally advanced inoperable or metastatic BC including at least 1 prior line of hormonal therapy in combination with an approved CDK4/6 inhibitor
6. Have no known active or symptomatic central nervous system (CNS) disease
7. Eastern Cooperative Oncology Group Performance Status (ECOG PS) ≤ 2

Metastatic Castration-Resistant Prostate Cancer:

1. Diagnosis of metastatic castration-resistant prostate cancer with disease progression despite castrate levels of testosterone
2. Evidence of disease progression as determined by Investigator per standard criteria
3. Have no known active or symptomatic CNS disease
4. Received prior therapy with anti-androgen(s) and taxane-based chemotherapy for castration-resistant disease
5. ECOG PS ≤ 2

Key Exclusion Criteria for All Cohorts:

1. Have received chemotherapy, hormonal therapy (with the exception of ongoing LHRH analogs in male patients and premenopausal women), radiation, or biological anti-cancer therapy within 14 days prior to the first dose of NUV-422
2. Has a history of or current use of bevacizumab (glioma and brain metastases only)
3. Received treatment with an investigational agent for any indication within 14 days for non-myelosuppressive agent or 21 days (or < 5 half-lives) for myelosuppressive agent prior to the first dose of NUV-422
4. Requires systemic corticosteroid therapy > 4 mg/day (> 2 mg/day for Expansion Cohort 2) of dexamethasone or equivalent or increasing doses of systemic corticosteroids during the 7 days prior to enrollment
5. Requires anti-seizure medications that are known to be strong inducers of CYP3A4/5 enzymes (carbamazepine, phenytoin) or has a recent history of uncontrolled or intermittent seizures
6. Females who are pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Phase 1 Dose Escalation: Safety and tolerability of NUV-422 to determine the recommended Phase 2 dose (RP2D) | During the DLT period (28 days)
  Incidence of treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), and dose-limiting toxicities (DLTs)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Arizona Oncology Associates, Tucson, Arizona
  - Miami Cancer Institute, Miami, Florida
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Carolina BioOncology Institute, Huntersville, North Carolina
  - Prisma Health Cancer Institute, Greenville, South Carolina
  - Texas Oncology P.A. Austin, Austin, Texas
  - Texas Oncology-Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Texas Oncology, Tyler, Texas
  - University of Utah Huntsman Cancer Institute, Salt Lake City, Utah
  - Virginia Cancer Specialists, Fairfax, Virginia